CLINICAL TRIAL: NCT00328107
Title: Evaluation of the Immunogenicity and Safety of Two Preparations of Trivalent Recombinant Baculovirus-Expressed Hemagglutinin Influenza Vaccine Administered Intramuscularly in Healthy Adults Ages 18-49 Years.
Brief Title: Immunogenicity and Safety of Trivalent Recombinant Hemagglutinin Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Protein Sciences Corporation (Industry)
Responsible Party: Manon MJ Cox, Protein Sciences Corporation
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: PSC01
Record Dates: First submitted 2006-05-17; First posted 2006-05-19 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluBlok

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose (Experimental): Recombinant Trivalent Hemagglutinin Influenza Vaccine, 2004/05 formulation containing 45μg of each hemagglutinin derived from A/Wyoming/3/03(H3N2) and 15μg from A/New Caledonia/20/99(H1N1) and B/Jiangsu/10/03
  Interventions: Biological: Influenza Vaccine, recombinant Hemagglutinin
- Full Dose (Experimental): Recombinant Trivalent Hemagglutinin Influenza Vaccine, 2004/05 formulation containing 45μg of each hemagglutinin derived from A/Wyoming/3/03(H3N2), A/New Caledonia/20/99(H1N1) and B/Jiangsu/10/03
  Interventions: Biological: Influenza Vaccine, recombinant Hemagglutinin
- Placebo (Placebo Comparator): 0.9% Sodium Chloride
  Interventions: Biological: Influenza Vaccine, recombinant Hemagglutinin

INTERVENTIONS:
Biological: Influenza Vaccine, recombinant Hemagglutinin — 0.5mL dose for IM injection
  Other Names: FluBlok; rHA; rHA0; recombinant hemagglutinin

SUMMARY:
The purpose of this study was to determine the dose-related safety, immunogenicity, and protective efficacy of a trivalent recombinant hemagglutinin influenza vaccine in healthy adults.

DETAILED DESCRIPTION:
All currently licensed influenza vaccines in the United States are produced in embryonated hen's eggs. There are several well-recognized disadvantages to the use of eggs as the substrate for influenza vaccine. Eggs require specialized manufacturing facilities and could be difficult to scale up rapidly in response to an emerging need such as a pandemic. It is usually necessary to adapt candidate vaccine viruses for high-yield growth in eggs, a process that can be time consuming, is not always successful, and can select receptor variants that may have suboptimal immunogenicity. In addition, agricultural diseases that affect chicken flocks, and that might be an important issue in a pandemic due to an avian influenza virus strain, could easily disrupt the supply of eggs for vaccine manufacturing. Therefore, development of alternative substrates for influenza vaccine production has been identified as a high-priority objective.

One potential alternative method for production of influenza vaccine is expression of the influenza virus hemagglutinin (HA) using recombinant DNA techniques. This alternative avoids dependence on eggs and is very efficient because of the high levels of protein expression under the control of the baculovirus polyhedrin promoter.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable adults, aged 18-49 years.
* Provided informed consent prior to any study procedures.
* Able to comply with all study procedures.
* Available for follow-up for the duration of the influenza season.
* Women of child-bearing potential had a negative urine pregnancy test at the time of randomization and were willing to use an adequate form of contraception during the course of the study.

Exclusion Criteria:

* Any history of immunodeficiency or treatment with immunosuppressive medications. (Use of inhaled steroids or of topical steroids was not considered immunosuppressive; receipt of systemic glucocorticosteroids was not allowed if daily intake was >10 mg of prednisone or equivalent).
* Presence of high-risk conditions or other characteristics considered to be indications for influenza vaccination, as defined by the Advisory Committee on Immunization Practices (ACIP).
* Acute febrile illness (defined as having a temperature ≥100degreesF) or upper respiratory tract illness within 72 hours of vaccination.
* Use of experimental vaccines or any influenza vaccine after May 31st 2004 for the 2005 Southern Hemisphere or 2004 to 2005 Northern hemisphere epidemic seasons.
* Use of any experimental medication within 30 days prior to study vaccination
* Women who were pregnant or breast-feeding.
* Subjects with a history of Guillain-Barré syndrome.
* Receipt of parenteral immunoglobulin within 30 days prior to study vaccination.
* Any acute or chronic condition that, in the opinion of the investigator, would render vaccination unsafe or interfere with the evaluation of response.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 459 (Actual)
Dates: Start 2004-11; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and reactogenicity of trivalent recombinant hemagglutinin influenza vaccine in healthy adults aged 18-49 years | influenza season

SECONDARY OUTCOMES:
Evaluation of the protective efficacy of a trivalent recombinant hemagglutinin influenza vaccine at two different formulations in healthy adults aged 18-49 years | influenza season
Evaluation of the immunogenicity of the H1 and B components when formulated at either 15μg or 45μg per component in healthy adults aged 18-49 years | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: John Treanor, MD, Principal Investigator — University of Rochester
Locations (3):
- United States (3):
  - Rochester Medical Center, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Virginia Health System, Charlottesville, Virginia

REFERENCES:
- [Result] Treanor JJ, Schiff GM, Hayden FG, Brady RC, Hay CM, Meyer AL, Holden-Wiltse J, Liang H, Gilbert A, Cox M. Safety and immunogenicity of a baculovirus-expressed hemagglutinin influenza vaccine: a randomized controlled trial. JAMA. 2007 Apr 11;297(14):1577-82. doi: 10.1001/jama.297.14.1577. PMID 17426277
- See also: Related Info — http://proteinsciences.com